CLINICAL TRIAL: NCT04516460
Title: Efficacy of PuraStat for the Prevention of Delayed Bleeding After Endoscopic Resection of Colorectal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Pedro Hispano (Other)
Responsible Party: Principal Investigator, Francisco Baldaque Silva, Principal Investigator, Hospital Pedro Hispano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 52/20/RS
Record Dates: First submitted 2020-07-28; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Bleeding After Resection of Colorectal Neoplastic Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PuraStat (Experimental): Interventional arm: PuraStat® applied through a catheter delivery system via the endoscope is used to prevent bleeding after endoscopic resection
  Interventions: Device: Interventional arm: endoscopic resection plus PuraStat®

INTERVENTIONS:
Device: Interventional arm: endoscopic resection plus PuraStat® — Interventional arm: PuraStat® applied through a catheter delivery system via the endoscope is used to prevent bleeding after endoscopic resection of colorectal neoplastic lesions

SUMMARY:
A Prospective Interventional Multicentric Study to Evaluate Effectiveness and Safety of PuraStat in the Management of delayed bleeding following Endoscopic Mucosal Resection (EMR) in the colon and rectum.

DETAILED DESCRIPTION:
1. BACKGROUND & RATIONALE

   Endoscopic resection is used frequently for the management of benign and early neoplastic gastrointestinal (GI) lesions. Bleeding can occur during or after endoscopic mucosal resection and may impact patient's morbidity and mortality. Following colorectal endoscopic mucosal resection (EMR), the delayed bleeding rate may range between 5 and 9% [1, 2]. Several endoscopic hemostatic therapies based on coagulation, clipping or adrenaline may be used to prevent or treat post-polypectomy bleeding.

   Adrenaline has a temporary effect, is associated with reduction of early post-polypectomy bleeding but does not reduce the risk of delayed bleeding [3]. The use of coagulation forceps may be associated with complications such as perforation [4] and necrosis [5], and its role on the prevention of delayed bleeding is not established yet [3]. Different hemoclips may be applied in this context. However, their use may be technically difficult in some colonic areas and may be more difficult to deploy and to remain in place for long periods in the left colon and rectum where the colonic wall is thicker [6]. Clips are effective in complete closure of mucosal defects in only 57% of cases [7] [6] and that has impact on the prevention of delayed bleeding. Most of the studies evaluating theses different strategies are performed in high-volume centers with high expertise on endoscopic therapy.

   There is a need for a safe, effective and friendly to use preventive hemostatic therapy, that would be easier to deploy, irrespective of mucosal defect size, location and endoscopist's expertise.

   PuraStat is a synthetic self-assembling aqueous peptide that ionises rapidly to form a network of nanofibers when it comes into contact with blood or ionic fluid. It is a safe, non-biogenic, biocompatible, resorbable peptide hydrogel with no infection transmission risk and is available in 1ml, 3ml and 5ml syringes. The syringe is connected to a dedicated endoscopy catheter that is placed through the working channel of the endoscope. It is CE marked and indicated for use for haemostasis in the following situations encountered, during surgery, when haemostasis by ligation or standard means is insufficient or impractical: bleeding from small blood vessels and oozing from capillaries of the parenchyma of solid organs, oozing from vascular anastomoses, bleeding from small blood vessels and oozing from capillaries of the GI tract following surgical procedures. PuraStat is also indicated for the reduction of delayed bleeding following gastrointestinal endoscopic submucosal dissection (ESD) procedures in the colon.

   Studies have suggested that PuraStat may have a wide range of benefits, including haemostasis and regeneration of soft tissues [8-18].

   A 25-patient study in cardiovascular surgery with PuraStat showed that no postoperative bleeding or adverse events [8]. Ohri et al.2018, published a 50 patient feasibility and efficacy study in adult cardiac surgery, concluding PuraStat as easy-to-use and effective haemostatic agent in a wide range of cardiac procedures [9]. In Addition Ananda et al, 2017 undertook a 60 patient haemostatic efficacy and feasibility study in ENT turbinate surgery with no nasal packing demonstrating in all patients there was no post-operative re-bleeding observed and healing went well in absence of adhesion formation[10] . A 12-patient GI pilot study assessed PuraStat's haemostatic efficacy following endoscopic resection of gastric neoplasia was conducted and PuraStat was found to be effective [15]. Pioche et al. in 2016 performed a study of PuraStat used prophylactically following endoscopic resection in patients of high risk of delayed bleeding, demonstrating a delayed bleeding rate of 6.2% [16]. Uraoka et al. demonstrated the use of PuraStat for preventing delayed bleeding and enhancing gastric ulcer healing following ESD with good effect [17]. Most recently in 2018 a study was published by Bhandari et al. where PuraStat was used on 100 patients undergoing endoscopic resection to assess safety, feasibility, haemostatic efficacy and delayed bleeding rates. This study showed PuraStat to be effective at controlling bleeding and a delayed bleeding rate of 3% [18].

   PuraStat is a novel haemostatic agent with published haemostatic safety and efficacy data in a number of surgical / interventional areas. However, there is limited trial and observation data in relation to delayed bleeding following endoscopic resection.

   The investigators aim to evaluate PuraStat's clinical effectiveness, safety and technical feasibility in the prevention of post colorectal EMR delayed bleeding.
2. AIMS & OBJECTIVES

   To conduct a prospective interventional, multicenter study to evaluate the use of PuraStat for the prevention of delayed bleeding following colorectal EMR.

   2.1 Primary Objective

   • To assess the incidence of delayed bleeding after colorectal EMR using PuraStat (definition above).

   2.2 Secondary Objectives
   * To assess the technical feasibility and ease of use of PuraStat when used in the prevention of GI bleeding
   * To monitor any unexpected reactions that may be attributed to the use of PuraStat
   * To evaluate the incidence of overall serious adverse events such as post-polypectomy syndrome, fever, pain or perforation.
3. STUDY DESIGN

   3.1 Summary of Study Design This is a prospective interventional, multicentric study to collect data on the clinical effectiveness, safety and feasibility of PuraStat in the prevention of delayed bleeding following colorectal EMR.

   3.2 Primary and Secondary Endpoints/Outcome Measures

   Primary Endpoint - Clinically relevant delayed bleeding rate (as defined above) Secondary Endpoints

   - Technical feasibility of PuraStat application to the desired site
   * Duration of application of PuraStat
   * Occurrence of Suspected Unexpected Serious Adverse Reactions (SUSAR) related to PuraStat
4. STUDY PARTICIPANTS 4.1 Study Setting

The research will be conducted across multiple participating sites with Hospital Pedro Hispano, Matosinhos, Portugal, acting as the sponsor

Sites:

1. Hospital Pedro Hispano, Matosinhos, Portugal
2. UZ Leuven (Leuven)
3. Karolinska University Hospital (Stockholm)

4.2 Overall Description of Study Participants

Patients will fall into the below category:

1. Those requiring prophylactic measures to prevent future GI bleeding after a high-risk endoscopic resection:

   Colorectal nonpedunculated lesions > 2cm

   4.3 Eligibility Criteria Inclusion Criteria

   All of the following:
   * Presence of 1 lesion >2cm in the colon or rectum
   * Patients able to give informed consent.
   * Patients over 18 years of age. Exclusion Criteria

   ANY of the following:

   • resection of more than one large (≥20mm) polyp

   • ulcerated lesion (Paris III morphology)

   • lesions with invasive component

   • inflammatory bowel disease

   • poor health condition (American Society of Anesthesiologists class IV)

   • resection by endoscopic submucosal dissection

   • incomplete EMR

   • use of clips in the mucosal defect

   • previous attempts of endoscopic resection of the same lesion

   • suspected deep damage in the muscularis propria

   • coagulation disorder (international normalized ratio >1.5, platelets <50)
   * pregnancy

   Periprocedural management with antiplatelets or anticoagulants will be performed according to the ESGE guidelines [19].

   The "antiplatelet therapy" category included treatment with aspirin, clopidogrel, double antiplatelet therapy and other antiaggregant. Aspirin will not be discontinued, but thienopyridines will be routinely discontinued 5 to 7 days before EMR and reintroduced the day after the procedure. Anticoagulant therapy category includes treatment with acenocumarol or warfarin, nonvitamin K oral anticoagulants (NOACs) and bridging therapy with low molecular weight heparin. Acenocumarol or warfarin will be discontinued 5 days before the procedure. Bridging therapy with heparin will be used as recommended. Before the procedure, an international normalized ratio (INR) <1.5 will be confirmed in patients who received anticoagulation therapy. NOACs will discontinued 48 to 72 hours before EMR and restarted the day after EMR.

5.SAMPLING This study aims to investigate the use, effectiveness, feasibility and safety of PuraStat in reducing delayed bleeding following EMR in the colon. Delayed bleeding in the colon following EMR is recorded as being between 5-9%. This is a feasibility study where the investigators aim to include approximately 144 patients treated with PuraStat over a 12 month period period.

6. STUDY PROCEDURES A dedicated Case report form (CRF) to capture data points will be designed and made available to all participating centres. The CRF will contain all of the data needed for the study but no patient identifiable details. All endoscopists participating in the study will be trained in the use of PuraStat. Patients will be followed up for evidence of [clinically relevant] delayed bleeding.

Experienced senior endoscopists (>100 successful EMRs each) will perform the procedures using conventional or high definition white light endoscopes. The lesion size will be measured either with open forceps or with the longitudinal edge of an open snare. Injection- assisted EMR with lifting solution with indigo carmin/methylene blue will be performed according to the literature.

ERBE models (VIO-200, VIO-300 or VIO 3 will be used in the automatic controlled mode (Endocut-Q, ERBE Electromedizin®, Tübingen, Germany) Coagulation of submucosal vessels by means of snare tip coagulation, argon plasma coagulation or coagulation forceps will be performed when the endoscopist considered it necessary. If bleeding occur during the procedure (immediate bleeding), specific prophylactic measures on selective vessels will be carried out and recorded.

7.1 Recruitment The investigators anticipate that all participating centers will recruit 144 patients.

7.2 Screening and Enrolment Ideally, all patients meeting the inclusion criteria for the study will be approached for inclusion to avoid potential bias. Patients will be provided with information about the procedure in an appropriate time frame. Signed informed consent will be obtained prospectively from the patient for the use of their data for inclusion in the study.

7.3 Study Assessments A secure electronic database will be used for data entry. Post colonoscopy assessment will be performed at 7 and 30 days by an external assessor by telephone interview.

See below for sample of data points to be collected:

A. Pre-Endoscopy

* Patient demographics (age, sex)
* Co-morbidities (diabetes, renal failure, cardiorespiratory)
* Use of anticoagulants and antiplatelets and date stopped (if applicable) and bridge therapy (if applicable)
* ASA score
* Previous endoscopic treatment
* Type of endoscopic procedure
* Haemoglobin & urea (at baseline or on admission)
* Vital signs (blood pressure, pulse)

B. At endoscopy

- Date of procedure

* Mode of sedation (general anaesthesia, propofol, or conscious sedation)
* Endoscopy findings
* Time of start and finish of resection (indirect assessment of difficulty of resection)
* mL of saline for subepithelial lyfting
* Type and size of snare used
* Type of resection procedure (polypectomy, en bloc EMR, piecemeal EMR)
* Lesion size
* Lesion location
* Lesion morphology (e.g Paris classification, NICE classification)
* Size of resection base
* Residual lesion (Y/N)
* Adjunctive use of clips, APC or prophylactic coagulation
* Indication for PuraStat - as a prophylactic agent to prevent bleeding
* Amount of PuraStat used (mls) over resected area
* Length in time of Purastat application
* Ease of Application:
* Catheter blockage (Y/N)
* Completeness of coverage (% of bleeding area covered)
* Intraprocedural Complications

C. Post endoscopy

* Complications (up to 30 days) as defined above
* Delayed perforation (time, treatment, outcome)
* Delayed bleeding (time, treatment, outcome)
* Post polypectomy syndrome (time, treatment, outcome)
* Emergency surgery (time, treatment, outcome)
* Death
* Other serious adverse events (cardiac/respiratory) resulting in hospitalisation/interventional treatment (time, treatment, outcome)
* Length of hospital admission
* Follow up endoscopy findings (where applicable - e.g. for further management of rebleeding or delayed bleeding within 30 days of primary procedure where PuraStat was used)

7.4 Discontinuation/Withdrawal of Participants from Study Treatment Patients will be able to opt to withdraw their data from the database at a later stage if so desired.

7.5 Definition of End of Study Each patient is considered a study participant for 30 days following the initial use of PuraStat. The final study end date is 30 days after PuraStat is used in the last patient recruited.

8. INTERVENTIONS 8.1 Description of Study Intervention / Treatment This is an interventional study of PuraStat used prophylactically to reduce delayed bleeding following EMR in the colon <2cm.

PuraStat is supplied in a pre-filled syringe and is currently available in 1mL, 3mL and 5mL syringes. It is delivered via a dedicated catheter passed through the working channel (minimum 2.8mm diameter) of the endoscope. It is applied to in the mucosal defect under direct visualisation at the end of the EMR procedure, ensuring to cover the entire resected area.

9. ASSESSMENT OF SAFETY Where a complication occurs that has the characteristics of a Suspected Unexpected Serious Adverse Reaction, (i.e. related' - that is, it resulted from administration of any of the research procedures; and 'unexpected' - that is, the type of event is not listed in the manufacturers information as an expected occurrence, and is also Serious - i.e. results in death, is life threatening, requires hospitalization or prolonged hospitalization, persistent or significant disability/incapacity, congenital anomaly or other important medical event) sites will be asked to report this to the Chief Investigator and the Chief Investigator will in turn report this information to the manufacturer directly. The Chief Investigator will also assess whether the event should be reported to the local Regulatory Agency.

10. DATA HANDLING AND RECORD KEEPING 10.1 Data Collection Forms Data will be recorded onto a dedicated CFR following the initial endoscopy where PuraStat was used. The anonymised data form will then be entered onto a secure password protected electronic database with appropriate backup systems and security protocols in place. No patient identifiable data will be stored on the database. The data collection forms and electronic database will capture information on data described above on points 9.3 A-C.

10.2 Data Management

All data will be inserted in a e-CRF/paper CRF along the different steps of the process: previously and immediately after colonoscopy and during the follow-up.

Complications will be externally assessed by phone call or during a clinic visit at 7 and 30 days after the procedure and after review of medical records.

All serious adverse will be reported to and reviewed by a data safety monitoring board.

Each patient will have an identification code number that will enable anonymized storing of all data.

All data will be stored in an anonymized electronic password protected database that will be assessed by the one member of the research group and one external assessor (in each hospital).

11. DATA ANALYSIS Description of Analysis Populations

All data will be anonymized stored. An intention to treat analysis will be performed in all included all patients. The per protocol analysis will include the cases in which complete mucosal defect treatment with PuraStat is achieved.

12. ETHICS 12.1 Participant Confidentiality The study staff will ensure that the participants' anonymity is maintained. The participants will be identified only participant's code number on the CRF and any electronic database. All documents will be stored securely and only accessible by study staff and authorized personnel. The study will comply with the Data Protection Act which requires data to be anonymized as soon as it is practical to do so

12.2 Other Ethical Considerations This study will be carried out subject to approval by each Institution research ethics committee. It will be carried out in accordance with the Medicine for Human Use (Clinical Trial) regulations (2004), International Conference for Harmonisation of Good Clinical Practice (ICH GCP) guidelines and World Association Declaration of Helsinki (1964) and Scotland (2000) amendments.

Patient confidentiality will be maintained throughout. No information will be disclosed or reproduced through which patients could be identified. Should new relevant information arise from other studies on PuraStat (e.g on safety or efficacy profile), the Sponsor will review this and disseminate the information appropriately to study participants.

12.3 Declaration of Helsinki The study will be carried out in accordance with the Declaration of Helsinki (1964) and Scotland (2000) amendments.

13. FINANCING AND INSURANCE The device has a CE mark and is covered by product liability insurance from the company, the evidence of which can be provided upon request. There will be no excess treatment costs associated with the study as the haemostatic device will be provided free of charge for the purpose of the study by the manufacture, 3-D Matrix.

14. RESOURCES, EQUIPMENT AND PHYSICAL FACILITIES

All included centres have high volume of therapeutic endoscopy, namely on endoscopic mucosal resection in the colon and rectum.

All participant endoscopists have high expertise on EMR of colorectal lesions. All procedures will be performed with high-definition endoscopy, with lesions characterization. ERBE electrosurgical units will be used in all procedures as described above.

15. DISSEMINATION AND OUTCOME The analysis of the data will be presented at national and international conferences. Results will subsequently be published in peer reviewed scientific journals and disseminated to relevant patient groups.

ELIGIBILITY:
Inclusion Criteria:

All of the following:

* Presence of 1 lesion >2cm in the colon or rectum
* Patients able to give informed consent.
* Patients over 18 years of age.

Exclusion Criteria:

ANY of the following:

* resection of more than one large (≥20mm) polyp
* ulcerated lesion (Paris III morphology)
* lesions with invasive component
* inflammatory bowel disease
* poor health condition (American Society of Anesthesiologists class IV) resection by -endoscopic submucosal dissection
* incomplete EMR
* use of clips in the mucosal defect
* previous attempts of endoscopic resection of the same lesion suspected deep damage in the muscularis propria
* coagulation disorder (international normalized ratio >1.5, platelets <50) pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-01-28 (Estimated); Study Completion 2022-01-28 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant delayed bleeding rate | 1 month after procedure
  (as defined above)

SECONDARY OUTCOMES:
Technical feasibility of PuraStat application to the desired site | 1 day
  1-Possible to apply all desired Purastat, 2-Possible to apply some Purastat, 3- Not possible to apply purastat
Duration of application of PuraStat | 1 day
  secs
Occurrence of Suspected Unexpected Serious Adverse Reactions (SUSAR) related to PuraStat | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Masami Omae, MD, Study Chair — Karolinska Hospital
Locations (1):
- Hospital Pedro Hispano, Matosinhos Municipality, Portugal